CLINICAL TRIAL: NCT05190770
Title: A Randomized Phase II Double-Blinded Study of The Efficacy of Oleogel-S10 (AP101) Gel for the Treatment of Grade 2/3 Radiation Dermatitis in Breast Cancer Patients
Brief Title: A Study of Oleogel-S10 Gel for the Treatment of Radiation Dermatitis in People With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21-091
Record Dates: First submitted 2021-12-29; First posted 2022-01-13 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Breast Cancer Stage; Breast Cancer Stage I; Breast Cancer Stage II; Breast Cancer Stage III; Breast Cancer Stage IV
Keywords: Radiation Dermatitis; PMRT; Breast cancer; Oleogel-S10; Triamcinolone acetonide; Memorial Sloan Kettering Cancer Center; 21-091
MeSH Terms: conditions — Breast Neoplasms; Radiodermatitis | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Triamcinolone + Oleogel-S10 (Experimental): 25 participants will be randomized to triamcinolone 0.1% cream once every morning and topical Oleogel-S10 gel once prior to bedtime for a 3 week period.
  Interventions: Drug: Triamcinolone Acetonide; Drug: Oleogel-S10
- Triamcinolone + Placebo (Placebo Comparator): 25 patients with breast cancer will be randomized to triamcinolone 0.1% cream once every morning (QAM) and vehicle gel once prior to bedtime for a 3 week period.
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Triamcinolone Acetonide — Triamcinolone acetonide is a derivative of prednisolone with high glucocorticoid activity and low mineralocorticoid activity. It is applied topically.
Drug: Oleogel-S10 — Oleogel-S10 consists of birch bark extract (TE): 10 mg/100 mg; Sunflower oil, refined: 90 mg/100 mg. It is applied topically.
  Arms: Triamcinolone + Oleogel-S10

SUMMARY:
The purpose of this study is find out whether Oleogel-S10 is an effective treatment for radiation dermatitis when it is used in combination with a standard wound treatment cream called triamcinolone. Oleogel-S10 has shortened the healing time for other types of skin wounds such as burns. Triamcinolone is a cream that is frequently used to treat moderate to severe skin conditions such as skin irritation caused by poison ivy, eczema, sunburn, and rashes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are receiving PMRT to the chest wall or post-lumpectomy RT to the whole breast cancer of any stage
* Age ≥ 18 years
* Patients who develop ARD grade 2/3 after fraction day 20 (when receiving 25 total fractions) or after fraction day 25 when receiving (30 total fraction inclusive of a 5 fraction boost) of radiation therapy with all locations of desquamation
* Able to self-administer topical interventions or provide for another person to apply the topical intervention
* Patients may be started on any topicals prior to study enrollment. Once patient is enrolled on study (on or before Day 1), patient must be able to discontinue other topicals (including topical steroids, Silvadene, calcineurin inhibitors) to the treatment area
* Patients have completed surgery or chemotherapy ≥ 4 weeks prior to start of radiation therapy. Patients may receive antibody-drug conjugates at any time before/during/after study
* Women of childbearing potential (WCBP) must have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Baseline (Day 0) and documented monthly.
* WCBP must agree to abstrain from sex or use a highly effective method of birth control* from the time of consent through visit 5.

  * Adequate contraceptive methods include those with a low failure rate, i.e., less than 1% per year, when used consistently and correctly, such as abstinence from sexual intercourse, and some double barrier methods (condom with spermicide) in conjunction with use by the partner of an intrauterine device, diaphragm with spermicide, oral contraceptives, birth control patch or vaginal ring, or injectable or implanted contraceptives. Abstinence is acceptable only as true abstinence: when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

A woman that is postmenopausal (≥2 years since last menstrual period) or permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy) is not considered a WCBP.

Exclusion Criteria:

* Patients who are receiving radiation therapy for inflammatory breast cancer or malignant fungating wound
* Known history of allergy to any ingredient of the study medication
* Patients with collagen-vascular disease/vasculitis
* Patients receiving hypofractionated radiation therapy
* Special populations:

  * patients who, in the opinion of the investigator have a condition that precludes their ability to provide an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alina Markova, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Memorial Sloan Kettering at Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Triamcinolone + Oleogel-S10 | Triamcinolone + Placebo
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Triamcinolone + Oleogel-S10 | Triamcinolone + Placebo | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Median (Full Range); unit: years] | 42 [28 to 72] | 56 [34 to 69] | 47 [28 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 8 | 9 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 9 | 17
  United Kingdom | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Wound Surface Area Reduction of Radiation Dermatitis Grade 2-3 Wound Size From Baseline to Day 14 (+/- 3 Days)
Description: The primary outcome of this study is the efficacy of Oleogel-S10 in reducing radiation dermatitis grade 2-3 wound size in patient with breast cancer undergoing external beam radiation therapy. Clinical assessment at all study visits, including wound surface area and adverse events will be performed by a dermatologist. Wound size will be measured using a HIPAA compliant 3D clinical imaging system.
Time Frame: 14 days from baseline (+/- 3 days)
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Triamcinolone + Oleogel-S10 | Triamcinolone + Placebo
Number analyzed (Participants) | 9 | 9
cm^2
  Baseline | 10.3 (16.8) | 25.3 (65.2)
  Day 14 | 0.5 (0.8) | 4.1 (10.0)

ADVERSE EVENTS:
Time Frame: 14 days from baseline
Arm/Group | Triamcinolone + Oleogel-S10 | Triamcinolone + Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 3/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Triamcinolone + Oleogel-S10 (N=9) | Triamcinolone + Placebo (N=9)
Skin infection (Infections and infestations) | 2 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-13): https://cdn.clinicaltrials.gov/large-docs/70/NCT05190770/Prot_SAP_000.pdf